CLINICAL TRIAL: NCT00598819
Title: A Prospective Study With a New Device for the Monitoring of Cerebral Oxygenation on Healthy Volunteers
Brief Title: A Prospective Study of a New Device for Monitoring Cerebral Oxygenation on Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Jeffrey Milliken, MD, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-5593
Record Dates: First submitted 2007-12-19; First posted 2008-01-23 (Estimated); Results first posted 2010-07-07 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-08

CONDITIONS: Cerebral Ischemia
Keywords: Cerebral Oxygenation; Oxygen Monitoring
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy Volunteers (Experimental): Healthy subjects testing the device.
  Interventions: Device: CDI 1000 COM

INTERVENTIONS:
Device: CDI 1000 COM — CDI 1000 COM sensors were attached to subject's forehead for a 12 hour period.
  Other Names: Terumo CDI 1000 COM

SUMMARY:
The purpose of this study is to determine whether a new cerebral oxygen monitoring device is effective and comparatively similar to the current approved devices.

DETAILED DESCRIPTION:
Cerebral oxygenation monitoring is an innovative way to monitoring cardiac surgery patients intraoperatively to reduce the incidence of postoperative hypoxic side effects. There are a number of approved devices already in the market that have proved their effectivity.

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy male or Female Volunteers
* 18 years old or older
* Capable and willing to operate a bicycle
* Understand enough about the risks and benefits of the study to be able to make an informed decision before agreeing to be in the study

EXLUSION CRITERIA:

* History of Cerebrovascular Disease
* History of Skin Problems on Forehead (Skin Rashes, Acne, Allergies, etc.)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey C Milliken, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy Volunteers
Pre-assignment Details: Physical Exam to confirm healthy status. The physical exam was performed by the investigator that is a licensed Medical Doctor.
Groups:
- Healthy Volunteers: The participants were young adults (18 year-old or Older) who met the inclusion/exclusion criteria for the study and passed a physical exam. Subjects were fitted with the device, and laid down for 4 hours, sat upright for 30 minutes and rode an exercise bicycle for 30-45 minutes. The physical exam and device fitting was performed by the investigator.
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Harm to Skin From Attachment of Sensor to Forehead: Cuts, Bruising, Rash or Allergic Reactions to Adhesive.
Description: Measurement of reactions to the sensor's attachment to the skin on the forehead. Measurement of the outcome is either reaction or no reaction. This means that all subjects are either measured as having a reaction at all or having no reaction at all. Measurement and reactions assessment performed by the investigator.
Time Frame: attachment of sensor to 24 hours post-removal
Population: The number of participants was determined by protocol specifications.
Measure: Number; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 14
Participants
  Harm caused by sensor | 0
  No harm caused by sensor | 14

2. Primary Outcome: Overheating of Skin Underneath Sensor.
Description: The Principal measure for this outcome was discomfort and potential harm from overheating while attached to an active study participant. The investigator of the study asked to the participant if he/she felt:
  • Discomfort in the sensor application zone; Itching, Burning sensation and/or Pain. The skin was examined before and after the sensor application. All the assessments were performed by the principal investigator of the study.
Time Frame: placement of sensor to 10 minutes post-removal.
Measure: Number; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 14
Participants
  Overheating underneath sensor | 0
  No overheating underneath sensor | 14

3. Secondary Outcome: Sensor Fits Well on Subjects Forehead
Description: How well the sensor seems to fit on the subject's forehead in terms of curvature, comfort and adherence. The fitting assessment was assessed visually and determined based in the size of the sensor and the length of forehead covered, also the adhesion test was performed by hanging weight of 2 LBS on the sensor for 10 min, recording if the sensor kept attached to the skin or not. All tests and measures were assessed by the investigator. All the characteristics of the sensor (curvature, comfort and adherence) were recorded on each subjects as "yes" or "no".
Time Frame: placement of sensor to end of study observation
Measure: Number; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 14
Participants
  Sensor fit well | 14
  Sensor did not fit well | 0

4. Secondary Outcome: Sensor Attachment Under Stress
Description: as for outcome 2
Time Frame: addition of stress on sensor to removal.
Measure: Number; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 14
Participants
  Sensor gave out under stress | 0
  Sensor held up to stress | 14

5. Primary Outcome: Overheating of Skin Underneath Sensor
Description: as for outcome 2
Time Frame: placement of sensor to immediately post-removal
Measure: Number; unit: Participants
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 14
Participants
  Overheating underneath sensor | 0
  No overheating underneath sensor | 14

ADVERSE EVENTS:
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
No Adverse Events (AE's) or Serious Adverse Events (SAE's) were reported in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less